CLINICAL TRIAL: NCT02672449
Title: Carbon Ions Boost Followed by Pelvic Photon Radiotherapy for High Risk Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: European Institute of Oncology (Other)
Collaborators: Associazione Italiana per la Ricerca sul Cancro (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEO 98
Record Dates: First submitted 2016-01-12; First posted 2016-02-03 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Adenocarcinoma of Prostate
Keywords: Prostate cancer; Carbon ions; Radiobiology; Radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- External beam radiotherapy (Experimental): A total of 65 consecutive newly diagnosed prostate cancer patients with 2013 NCCN high risk category will be consecutively enrolled in a prospective phase II trial on Carbon Ions Boost Followed by Pelvic Photon Radiotherapy .
  Interventions: Radiation: Carbon Ions Boost Followed by Pelvic Photon Radiotherapy

INTERVENTIONS:
Radiation: Carbon Ions Boost Followed by Pelvic Photon Radiotherapy — The patients will be enrolled either at the Centro Nazionale di Adroterapia Oncologica (CNAO), Pavia, Italy, at the Division of Radiation Oncology of the European Institute of Oncology (IEO), Milan, Italy, or at the Fondazione IRCCS Istituto Nazionale Tumori (INT), Milan, Italy. The treatment will include a boost phase on the whole prostate with carbon ions performed at CNAO followed by a pelvic photon RT, with IMRT performed with conventional fractionation of 1.8 Gy per fraction up to 45 Gy to the pelvic lymph nodes, prostate and seminal vesicles. The total dose prescribed to the prostate boost with carbon ions will be of 16.6 GyE in 4 fractions (4.15 GyE/fraction).

SUMMARY:
The aim of this research project is to test the feasibility and safety of a new treatment schedule for high risk prostate cancer that allows the administration of high doses to the prostate tumor with a mixed beam approach of carbon ions boost followed by pelvic IMRT.

DETAILED DESCRIPTION:
The present research project aims to improve the current treatment for high risk prostate cancer, evaluating the safety and feasibility of a new RT scheme of a carbon ions boost followed by pelvic photon RT.

A total of 65 consecutive patients will be enrolled in a prospective phase II trial. The patients will be enrolled either at Centro Nazionale di Adroterapia Oncologica (CNAO), Pavia, Italy, at the Division of Radiation Oncology of the European Institute of Oncology (IEO), Milan, Italy, or at the Fondazione IRCCS Istituto Nazionale Tumori (INT), Milan, Italy.

The treatment will include a boost phase on the whole prostate with carbon ions performed at CNAO followed by a pelvic photon IMRT performed with conventional fractionation of 1.8 Gy per fraction up to 45 Gy to the pelvic lymph nodes, prostate and seminal vesicles. All the patient data will be collected in a common database accessible from the 3 Institutions.

At CNAO, carbon ions beam is available for patient treatment since 2011. In comparison to the Japanese Center NIRS, the facility relies on active beam delivery using the rasterscan technique, which offers not only physical advantages with better sparing of normal tissues in the entrance channel, but also enables biologic plan optimization. The facility has the same equipment as the Carbon Ion Treatment Center in Heidelberg, Germany. At CNAO, 3D - 4D patient target localization is verified at each fraction by integrating orthogonal X-ray images and 3D real time optical tracking system.

At IEO and INT, the IMRT phase will be performed with the same treatment modality: volumetric-IMRT RapidArc by Varian Trilogy (IEO) and Varian DHX (INT) linacs, Varian Medical Systems, Palo Alto, CA, USA, with treatment based on the isocentric beam delivery, and pre-treatment image guidance for patient alignment via cone beam CT or portal imaging.

In phantom, quality assurance (QA) of each treatment will be performed before patient RT, in order to verify the consistency between calculated and delivered dose.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate, high-risk category according to NCCN version 2013 (T3a and/or PSA > 20 ng/ml and/or Gleason score of 8-10)
* cN0 and cM0
* Good performance status (ECOG<2)
* No previous pelvic RT
* No previous prostatectomy
* No concomitant bowel inflammatory disease or other serious comorbidities
* Good urinary flow (peak flow > 10 ml/s)
* No previous invasive cancer (within 5 years before the PCa diagnosis) apart from non-melanoma skin malignancies.

Exclusion criteria

* Pelvic lymph node metastasis (N1)
* Distant metastasis (M1)
* Urinary obstructive symptoms (IPSS > 20)
* Previous pelvic radiotherapy
* Severe systemic disorders
* Concomitant disorders including: chronic urinary or intestinal inflammatory conditions (for example, ulcerous recto-colitis, Crohn disease), anti-coagulant treatment (warfarin, heparin)
* Previous malignancy except for skin non-melanoma cancer or 3-year disease free interval from previous malignancy like in situ cervix cancer or non muscle invasive bladder cancer
* Non conformity of the radiotherapy dose distribution when compared to the dose constraints
* Psychiatric disorders or any other condition that can can make unreliable the informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Grade 3 or Grade 4 adverse events that are related to radiotherapy treatment according to the validated scale Radiotherapy Oncology Group / European Organization for Research and Treatment of Cancer (RTOG / EORTC). | one month after radiotherapy
  Toxicity and quality of life data will be prospectively assessed and analysed descriptively. Toxicities will be graded according to the Common Toxicity Criteria for adverse events (CTCAE) toxicity criteria v4.0 and Radiotherapy Oncology Group/European Organization for Research and Treatment of Cancer (RTOG/EORTC) criteria. Inacceptable toxicity will be > 3 patients with acute side effects grade 4, or > 3 patients with late RTOG/EORTC, CTCAE side effects grade 4, or > 3 patients with late RTOG/EORTC, CTCAE side effects grade 3, or any grade 5 toxicity.

SECONDARY OUTCOMES:
Number of patients who experienced late toxicity with Grade 3 or Grade 4 adverse events according to Scala CTCAE v4.0 toxicity criteria and scale RTOG / EORTC | two years
Number of patients with biochemical progression free survival measuring the PSA level | two years
  Biochemical progression free survival will be measured from the beginning date of RT to the date of PSA elevation. PSA relapse is defined according to the Consensus Statement of the American Society of Radiation Oncology (ASTRO) as elevation of PSA levels nadir + 2 ng/ml and confirmed by one measurement
Number of patients who experienced local or distance recurrence of disease assessed through radiological controls (Choline PET Scan, MRI) | two years
  It will be considered pattern of failure relapse in the same prostate lobe, in other lobes, in lymph nodes, in other distant sites.
Overall survival assessed by number of patients alive (with or without relapse) after the treatment | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Orecchia, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of oncology, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marvaso G, Jereczek-Fossa BA, Riva G, Bassi C, Fodor C, Ciardo D, Cambria R, Pansini F, Zerini D, De Marco P, Cattani F, De Cobelli O, Orecchia R. High-Risk Prostate Cancer and Radiotherapy: The Past and the Future. A Benchmark for a New Mixed Beam Radiotherapy Approach. Clin Genitourin Cancer. 2017 Jun;15(3):376-383. doi: 10.1016/j.clgc.2017.01.007. Epub 2017 Jan 18. PMID 28190704
- [Derived] Jereczek-Fossa BA, Fanetti G, Fodor C, Ciardo D, Santoro L, Francia CM, Muto M, Surgo A, Zerini D, Marvaso G, Timon G, Romanelli P, Rondi E, Comi S, Cattani F, Golino F, Mazza S, Matei DV, Ferro M, Musi G, Nole F, de Cobelli O, Ost P, Orecchia R. Salvage Stereotactic Body Radiotherapy for Isolated Lymph Node Recurrent Prostate Cancer: Single Institution Series of 94 Consecutive Patients and 124 Lymph Nodes. Clin Genitourin Cancer. 2017 Aug;15(4):e623-e632. doi: 10.1016/j.clgc.2017.01.004. Epub 2017 Jan 11. PMID 28185875